CLINICAL TRIAL: NCT00579709
Title: Thymus Transplantation With Immunosuppression, #884
Brief Title: Thymus Transplantation With Immunosuppression
Acronym: 884
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013734; R01AI047040 (NIH); R01AI054843 (NIH); 3R56AI047040-11A1S1 (NIH); R56 Bridge R01AI4704011A1 (Other: NIH American Recovery and Reinvestment Act (ARRA) of 2009); 2R01AI047040-11A2 (NIH); 5K12HD043494-09 (NIH); #884
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: DiGeorge Syndrome; DiGeorge Anomaly; Complete DiGeorge Anomaly; Complete DiGeorge Syndrome
Keywords: Thymus Transplantation; DiGeorge Anomaly; DiGeorge Syndrome; Athymia; Low T cell numbers; Immunoreconstitution; Immunodeficiency; Complete DiGeorge; Typical DiGeorge; Atypical DiGeorge; Complete DiGeorge Anomaly
MeSH Terms: conditions — DiGeorge Syndrome; Thymic aplasia; Immunologic Deficiency Syndromes | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Thymus Tissue for Transplantation
  Interventions: Biological: Thymus Tissue for Transplantation

INTERVENTIONS:
Biological: Thymus Tissue for Transplantation — 3 Thymoglobulin doses given prior to thymus tx. Atypical subjects given Cyclosporine (Csa) pre-tx. Desired Csa concentration 180-300ng/ml. If post-tx T cell count remained <4000/cumm Csa weaned over 8 weeks. If T cell >4,000/cumm, Csa held at 180-300ng/ml.
  Thymus tissue, donor, & mother of donor were screened for transplant safety. In operating room, thymic slices were transplanted into quadriceps muscle in 1 or both legs.
  Subjects had routine blood research immune evaluations. 2-3 months post-tx, open biopsy of allograft. Immune blood studies continued on surviving subjects until January 2010. Biological Mother: Mother provided blood sample used for DNA extraction, to identify/look for maternal T cell presence in recipient pre-tx, and/or for immune testing post-tx.
  Other Names: IND 9836; Thymus Tissue Transplant

SUMMARY:
The research purpose is to determine if thymus transplantation with immunosuppression is a safe and effective treatment for complete DiGeorge anomaly. The research includes studies to evaluate whether thymus transplantation results in complete DiGeorge anomaly subjects developing a normal immune system.

DETAILED DESCRIPTION:
DiGeorge anomaly is a complex of cardiac defects, parathyroid deficiency, and thymus absence, resulting in profound T-cell deficiency. There is a spectrum of disease in DiGeorge anomaly with respect to all three defects. For complete DiGeorge anomaly subjects with severe T cell defect, the PI had shown that thymus transplantation is safe and efficacious without pretransplantation immunosuppression and with pretransplantation Thymoglobulin and cyclosporine.

Some DiGeorge patients have very poor T cell function and are at risk of death from infection or other immune problems; however, these patients have enough T cell function to reject grafts. This protocol was designed for these patients. Atypical phenotype and some typical phenotype DiGeorge subjects were included in this protocol.

Atypical complete DiGeorge anomaly patients have rash, lymphadenopathy, and oligoclonal T cell proliferations. The T cells have no markers of thymic function (they do not co-express CD45RA and CD62L; they do not contain T cell receptor rearrangement excision circles, TRECs).

Typical complete DiGeorge anomaly patients in this protocol are those whose PHA response >20 fold. Although these patients have very low T cell function, it may be enough to reject a transplant, so Thymoglobulin was used.

ELIGIBILITY:
Transplant Inclusion

* No age limit
* Thyroid studies must be done and if abnormal, must be on therapy

DiGeorge diagnosis - must have 1 symptom from the following list:

* Heart defect
* Hypocalcemia requiring replacement
* 22q11 hemizygosity
* 10p13 hemizygosity
* CHARGE association
* Abnormal ears plus mother with diabetes (type I, type II, or gestational)

Atypical Diagnosis:

* Must have, or have had, a rash. If rash present, biopsy of rash must show T cells in skin. If rash & adenopathy resolved, must still have oligoclonal T cells.
* Within 1 month of tx must have PHA response >20 fold above background or >5,000 cpm, whichever is higher, or response can be < this.
* Circulating CD3+ T cells >50/mm3 but CD45RA+CD62L+CD3+ T cells <50/mm or <5% of CD3 count, whichever is higher (must be done 2x)
* Immunoscope with >40% oligoclonal TCRBV families. A 2nd test per sponsor discretion if T cell numbers increase or activation status changes.
* If TREC done pre-tx must have TRECs <100 per 100,000 CD3+ cells.

Typical Diagnosis:

* Circulating CD3+ CD45RA+ CD62L+ T cells and <50/mm3 or <5% of total T cells
* PHA response >20 fold above background or >5,000 cpm, whichever is higher.
* 2 studies must show similar immunological findings qualify for this study.
* TRECs, if done, should be <100/100,000 CD3 cells

Transplant Exclusion:

* Heart surgery <4 weeks pre-tx date
* Heart surgery anticipated w/in 3 months of proposed tx
* Rejection by surgeon or anesthesiologist as surgical candidates
* Lack of sufficient muscle tissue to accept 0.2 grams/kg transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-07; Primary Completion 2006-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability of Thymoglobulin and cyclosporine followed by thymus transplantation: Survival at 1 year post-transplantation. | 1 year post-transplantation

SECONDARY OUTCOMES:
Use of additional post transplant immunosuppression after that listed in the protocol. | The post thymus transplantation period
  Use of additional post transplant immunosuppression after that listed in the protocol.
Allograft biopsy used to evaluate graft rejection | 2 to 4 months post-transplant
  Evidence of thymus allograft rejection by immunohistochemistry of biopsy
CD3 count | 10 - 14 months post-transplantation
  CD3 count in cells/mm3
Thymopoiesis | 2-4 months after thymus transplantation
  Evidence of thymopoiesis in thymus allograft by immunohistochemistry of a biopsy
CD4 count | 10-14 months after thymus transplantation
  CD4 count in cells/mm3
CD8 count | 10-14 months after thymus transplantation
  CD8 count in cells/mm3
naive CD4 count | 10-14 months after thymus transplantation
  naive CD4 count in cells/mm3
naive CD8 count | 10-14 months after thymus transplantation
  naive CD8 count in cells/mm3

CONTACTS AND LOCATIONS:
Overall Officials: M. Louise Markert, MD, PhD, Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Background] Chinn IK, Olson JA, Skinner MA, McCarthy EA, Gupton SE, Chen DF, Bonilla FA, Roberts RL, Kanariou MG, Devlin BH, Markert ML. Mechanisms of tolerance to parental parathyroid tissue when combined with human allogeneic thymus transplantation. J Allergy Clin Immunol. 2010 Oct;126(4):814-820.e8. doi: 10.1016/j.jaci.2010.07.016. Epub 2010 Sep 15. PMID 20832849
- [Result] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sedlak DA, Sempowski GD, Hale LP, Rice HE, Mahaffey SM, Skinner MA. Postnatal thymus transplantation with immunosuppression as treatment for DiGeorge syndrome. Blood. 2004 Oct 15;104(8):2574-81. doi: 10.1182/blood-2003-08-2984. Epub 2004 Apr 20. PMID 15100156
- [Result] Markert ML, Devlin BH, McCarthy EA. Thymus transplantation. Clin Immunol. 2010 May;135(2):236-46. doi: 10.1016/j.clim.2010.02.007. Epub 2010 Mar 16. PMID 20236866
- [Result] Markert ML and Devlin BH. Thymic reconstitution (in Rich RR, Shearer WT, Fleischer T, Schroeder HW, Weyand CM, Frew A, eds., Clinical Immunology 3rd edn., Elsevier, Edinburgh) p 1253-1262, 2008.
- [Result] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Result] Selim MA, Markert ML, Burchette JL, Herman CM, Turner JW. The cutaneous manifestations of atypical complete DiGeorge syndrome: a histopathologic and immunohistochemical study. J Cutan Pathol. 2008 Apr;35(4):380-5. doi: 10.1111/j.1600-0560.2007.00816.x. PMID 18333898
- [Result] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Result] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759
- [Result] Hudson LL, Louise Markert M, Devlin BH, Haynes BF, Sempowski GD. Human T cell reconstitution in DiGeorge syndrome and HIV-1 infection. Semin Immunol. 2007 Oct;19(5):297-309. doi: 10.1016/j.smim.2007.10.002. Epub 2007 Nov 26. PMID 18035553
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA, Li YJ. Factors affecting success of thymus transplantation for complete DiGeorge anomaly. Am J Transplant. 2008 Aug;8(8):1729-36. doi: 10.1111/j.1600-6143.2008.02301.x. Epub 2008 Jun 28. PMID 18557726
- [Result] Markert ML, Devlin BH, McCarthy EA, Chinn IK, Hale LP. Thymus Transplantation in Thymus Gland Pathology: Clinical, Diagnostic, and Therapeutic Features. Eds Lavinin C, Moran CA, Morandi U, Schoenhuber R. Springer-Verlag Italia, Milan, 2008, pp 255-267.
- [Result] Markert ML, Devlin BH, Chinn IK, McCarthy EA. Thymus transplantation in complete DiGeorge anomaly. Immunol Res. 2009;44(1-3):61-70. doi: 10.1007/s12026-008-8082-5. PMID 19066739
- [Result] Markert ML, Marques JG, Neven B, Devlin BH, McCarthy EA, Chinn IK, Albuquerque AS, Silva SL, Pignata C, de Saint Basile G, Victorino RM, Picard C, Debre M, Mahlaoui N, Fischer A, Sousa AE. First use of thymus transplantation therapy for FOXN1 deficiency (nude/SCID): a report of 2 cases. Blood. 2011 Jan 13;117(2):688-96. doi: 10.1182/blood-2010-06-292490. Epub 2010 Oct 26. PMID 20978268
- [Result] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sempowski GD, Rhein ME, Szabolcs P, Hale LP, Buckley RH, Coyne KE, Rice HE, Mahaffey SM, Skinner MA. Complete DiGeorge syndrome: development of rash, lymphadenopathy, and oligoclonal T cells in 5 cases. J Allergy Clin Immunol. 2004 Apr;113(4):734-41. doi: 10.1016/j.jaci.2004.01.766. PMID 15100681
- [Result] Albuquerque AS, Marques JG, Silva SL, Ligeiro D, Devlin BH, Dutrieux J, Cheynier R, Pignata C, Victorino RM, Markert ML, Sousa AE. Human FOXN1-deficiency is associated with alphabeta double-negative and FoxP3+ T-cell expansions that are distinctly modulated upon thymic transplantation. PLoS One. 2012;7(5):e37042. doi: 10.1371/journal.pone.0037042. Epub 2012 May 10. PMID 22590644
- [Result] Chinn IK, Milner JD, Scheinberg P, Douek DC, Markert ML. Thymus transplantation restores the repertoires of forkhead box protein 3 (FoxP3)+ and FoxP3- T cells in complete DiGeorge anomaly. Clin Exp Immunol. 2013 Jul;173(1):140-9. doi: 10.1111/cei.12088. PMID 23607606